CLINICAL TRIAL: NCT04944355
Title: Urinary Tract Injuries During Caesarean Section for Morbidly Adherent Placenta: Prospective and Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoy Kedes Roshdy Said, Urinary tract injuries during caesarean section for morbidly adherent placenta: prospective and retrospective study, Assiut University
Other Study IDs: Urinary tract injuries at MAP
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-04

CONDITIONS: Urinary Tract Injuries During Caesarean Section for Morbidly Adherent Placenta: Prospective and Retrospective Study
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasound — diagnosis of morbid adherent placenta and incidence of urinary tract injuries during surgery
  Other Names: doppler

SUMMARY:
M1- evaluates the cases of lower urinary tract injuries during caesarean section with or without hysterectomy in cases with morbid placental adherence in the period between years 2018 and 2021. This study was carried out in assiut university women health hospital M 2- Clarification of the risk factors and outcome of urinary tract injuries.

DETAILED DESCRIPTION:
Placenta accreta spectrum disorder (PAS), also called abnormally invasive placenta (AIP), describes a clinical situation where the placenta does not detach spontaneously after delivery and cannot be forcibly removed without causing massive and potentially life-threatening bleeding(1-2) The incidence of PAS is rising worldwide(3) PAS is one of the most dangerous conditions of the pregnancy as it is significantly associated with maternal morbidity and mortality.(4) PAS may occur after any kind of procedure that causes damage to the endometrium, including curettage, manual removal of the placenta, uterine-artery embolization, or myomectomy(5-6) a full thickness surgical scar is associated with both the absence of endometrial re-epithelialization and vascular remodelling around the scar area, and this may lead to abnormally invasive placentation (increta/percreta).(7) Ultrasound is the first-line imaging tool for the screening and diagnosis of PAS. However, it is now well-established that magnetic resonance imaging (MRI) has a role in the diagnosis of PAS, with high sensitivity and specificity(8-9) Urinary bladder injury is one of the operative morbidities of cesarean section. It occurs in 0.08% - 0.94% of cesarean sections(10) Repeated cesarean section and type of morbidly adherent placenta (MAP) are considered the major risk factors for urinary tract injuries during cesarean delivery(11) Urinary bladder injury complicates about 11.7% of cesarean sections in women with placenta accreta spectrum (PAS)(12) The presence of tough adhesions between the bladder and the lower uterine segment carries the risk of urinary bladder injury. Trial of separation of the bladder in such circumstances may result in bladder injury. Filling of the bladder will delineate the contour of the bladder and clarify the proper plane of dissection (13)

ELIGIBILITY:
Inclusion Criteria:

* All cases in the 3rd trimester admitted to Asyut university women health hospital and diagnosed antenatally as having morbidly adherent placenta

  * Confirmed diagnosis of MAP.
  * Peri partum hysterectomy for MAP.
  * Complicated CS without hysterectomy
  * Maternal age between 18 and 45 yrs
  * No other medical diseases

Exclusion Criteria:

* associated other uterine pathology
* Refusal of the patient
* Emergency CS before confirming MAP diagnosis.
* Urinary tract injuries due to other causes than MAP
* Presence of major medical disorders e.g. DM, PE, Cardiac lesion, Coagulopathy, liver diseases or kidney diseases
* Postpartum depression.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female
Study Population: 1. This cross-sectional study will be conducted in Assiut University Hospital by analysis of records of cesarian section with or without hysterectomy in patient with morbid adherent placenta will be conducted and the cases complicated by urinary tract injuries from october2018 to october 2021.
  2. The occurrence of urinary tract injuries will be estimated and the records of those with injuries will be analysed prospectively from October 2018 to october 2021and retrospectively in terms of site and characteristics of injury, difference in management by different specialists, requirement of urologist for management, type of suturing, need for cystoscopy and catheter in situ placement.
  Study design:
  This study is a prospective and retrospective study
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
• Evaluate the incidence of different types of lower urinary tract injuries during caesarean section with or without hysterectomy in cases with morbid placental adherence(bladder-ureteric-bladder and ureteric injuries) | BASELINE
  • Evaluate the incidence of different types of lower urinary tract injuries during caesarean section with or without hysterectomy in cases with morbid placental adherence(bladder-ureteric-bladder and ureteric injuries)

CONTACTS AND LOCATIONS:
Locations (1):
- Asyut university women health hospital, Asyut, Egypt

REFERENCES:
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899
- [Background] Chantraine F, Braun T, Gonser M, Henrich W, Tutschek B. Prenatal diagnosis of abnormally invasive placenta reduces maternal peripartum hemorrhage and morbidity. Acta Obstet Gynecol Scand. 2013 Apr;92(4):439-44. doi: 10.1111/aogs.12081. PMID 23331024
- [Background] Jauniaux E, Chantraine F, Silver RM, Langhoff-Roos J; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Epidemiology. Int J Gynaecol Obstet. 2018 Mar;140(3):265-273. doi: 10.1002/ijgo.12407. No abstract available. PMID 29405321
- [Background] Fitzpatrick KE, Sellers S, Spark P, Kurinczuk JJ, Brocklehurst P, Knight M. The management and outcomes of placenta accreta, increta, and percreta in the UK: a population-based descriptive study. BJOG. 2014 Jan;121(1):62-70; discussion 70-1. doi: 10.1111/1471-0528.12405. Epub 2013 Aug 7. PMID 23924326
- [Background] Silver RM, Branch DW. Placenta Accreta Spectrum. N Engl J Med. 2018 Apr 19;378(16):1529-1536. doi: 10.1056/NEJMcp1709324. No abstract available. PMID 29669225
- [Background] Baldwin HJ, Patterson JA, Nippita TA, Torvaldsen S, Ibiebele I, Simpson JM, Ford JB. Antecedents of Abnormally Invasive Placenta in Primiparous Women: Risk Associated With Gynecologic Procedures. Obstet Gynecol. 2018 Feb;131(2):227-233. doi: 10.1097/AOG.0000000000002434. PMID 29324602
- [Background] Jauniaux E, Bhide A. Prenatal ultrasound diagnosis and outcome of placenta previa accreta after cesarean delivery: a systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Jul;217(1):27-36. doi: 10.1016/j.ajog.2017.02.050. Epub 2017 Mar 6. PMID 28268196
- [Background] Familiari A, Liberati M, Lim P, Pagani G, Cali G, Buca D, Manzoli L, Flacco ME, Scambia G, D'antonio F. Diagnostic accuracy of magnetic resonance imaging in detecting the severity of abnormal invasive placenta: a systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2018 May;97(5):507-520. doi: 10.1111/aogs.13258. Epub 2017 Dec 13. PMID 29136274
- [Background] Morel O, Collins SL, Uzan-Augui J, Masselli G, Duan J, Chabot-Lecoanet AC, Braun T, Langhoff-Roos J, Soyer P, Chantraine F; International Society for Abnormally Invasive Placenta (IS-AIP). A proposal for standardized magnetic resonance imaging (MRI) descriptors of abnormally invasive placenta (AIP) - From the International Society for AIP. Diagn Interv Imaging. 2019 Jun;100(6):319-325. doi: 10.1016/j.diii.2019.02.004. Epub 2019 Mar 8. PMID 30853416
- [Background] Korniluk A, Kosinski P, Wielgos M. Intraoperative damage to the urinary bladder during cesarean section - literature review. Ginekol Pol. 2017;88(3):161-165. doi: 10.5603/GP.a2017.0031. No abstract available. PMID 28397207
- [Background] Salman L, Aharony S, Shmueli A, Wiznitzer A, Chen R, Gabbay-Benziv R. Urinary bladder injury during cesarean delivery: Maternal outcome from a contemporary large case series. Eur J Obstet Gynecol Reprod Biol. 2017 Jun;213:26-30. doi: 10.1016/j.ejogrb.2017.04.007. Epub 2017 Apr 5. PMID 28411456
- [Background] Alanwar A, Al-Sayed HM, Ibrahim AM, Elkotb AM, Abdelshafy A, Abdelhadi R, Abbas AM, Abdelmenam HS, Fares T, Nossair W, Abdallah AA, Sabaa H, Nawara M. Urinary tract injuries during cesarean section in patients with morbid placental adherence: retrospective cohort study. J Matern Fetal Neonatal Med. 2019 May;32(9):1461-1467. doi: 10.1080/14767058.2017.1408069. Epub 2017 Dec 3. PMID 29157027
- [Background] Ozcan HC, Balat O, Ugur MG, Sucu S, Tepe NB, Kazaz TG. Use of Bladder Filling to Prevent Urinary System Complications in the Management of Placenta Percreta: a Randomized Prospective Study. Geburtshilfe Frauenheilkd. 2018 Feb;78(2):173-178. doi: 10.1055/s-0044-100039. Epub 2018 Feb 19. PMID 29479114